CLINICAL TRIAL: NCT06567652
Title: Safety and Efficacy of Persistent Atrial Fibrillation Ablation With a Cryoballoon Technology
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Carlo de Asmundis, Head of the department: Heart Rhythm Management Centre, Postgraduate Course in Cardiac Electrophysiology and Pacing, Vrije Universiteit Brussel, Universitair Ziekenhuis, Universitair Ziekenhuis Brussel
Other Study IDs: PolarXpersistent
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: catheter ablation — All patients underwent pulmonary vein isolation (and eventually left atrial posterior wall isolation) with the POLARx™ cryoballoon system

SUMMARY:
The goal of this retrospective observational study is to learn about the safety and efficacy of cryoballoon catheter ablation in 80 patients with persistent atrial fibrillation using the PolarX (Boston scientific) cryoablation technology. The main question it aims to answer is if it is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* persistent atrial fibrillation patients undergoing first atrial fibrillation ablation procedure with PolarX cryoballoon

Exclusion Criteria:

* previous atrial fibrillation ablation or cardiac surgery,
* paroxysmal atrial fibrillation,
* congenital heart disease,
* non-treated coronary artery disease,
* intracavitary thrombus,
* significant valvular disease,
* contraindications to general anesthesia.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persistent atrial fibrillation patients undergoing first atrial fibrillation ablation procedure with PolarX cryoballoon
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness | 1 year follow-up
  Primary effectiveness failure is defined as the composite of any of the following occurrences:
  Failure to achieve acute procedural success at the index procedure (pulmonary vein isolation); More than one repeat procedure during the blanking period (within 90 days post-index procedure); Documented atrial fibrillation, or new onset of atrial flutter or atrial tachycardia event (≥ 30 seconds in duration or from a 10 second 12-lead ECG) Repeat procedure for atrial fibrillation, or new onset of atrial flutter or atrial tachycardia Electrical and/or pharmacological cardioversion
  • Prescribed a new antiarrhythmic drug not documented at baseline Prescribed a higher dose of antiarrhythmic drug documented at baseline
Safety of the procedure | The safety endpoint was evaluated at 7-days 30-days and 1-year follow-up
  Safety is defined as the composite of any of the following occurrences:
  Death Myocardial infarction Persistent gastroparesis/injury to vagus nerve Stroke/Transient ischemic attack Thromboembolism/ Air embolism Cardiac tamponade/perforation Pneumothorax Serious vascular access complications* Pulmonary edema/Heart Failure Ablation related atrioventricular block not attributable to medication effect or vasovagal reaction.
  Safety events (0-30 days post procedure) Symptomatic pericardial effusion Safety events (0-360 days post procedure) Atrial esophageal fistula Persistent Phrenic nerve injury Pulmonary Vein Stenosis
  * Including hematoma requiring intervention or prolongation of hospital stay, artero-venous fistulas or pseudoaneurysm.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel Heart Rhythm Management Center, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No